CLINICAL TRIAL: NCT01209143
Title: A Phase Ib, Open-Label, Pharmacokinetic Drug Interaction Study of the Hedgehog Pathway Inhibitor GDC-0449 in Combination With Rosiglitazone or Combined Oral Contraceptive in Patients With Locally Advanced or Metastatic Solid Tumors That Are Refractory to Standard Therapy or for Whom No Standard Therapy Exists
Brief Title: A Study of Pharmacokinetic Drug Interaction Study of the Hedgehog Pathway Inhibitor GDC-0449 in Combination With Rosiglitazone or Combined Oral Contraceptive in Patients With Locally Advanced or Metastatic Solid Tumors That Are Refractory to Standard Therapy or for Whom No Standard Therapy Exists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHH4593g; GO01353 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Solid Cancers
MeSH Terms: interventions — HhAntag691; Rosiglitazone; ovcon 35

ARMS (2):
- Vismodegib + rosiglitazone (Experimental): Participants received rosiglitazone 4 mg orally on Days 1 and 8 of the study. Participants also received vismodegib 150 mg orally once a day beginning on Day 2 until one of the following occurred; disease progression, intolerable toxicity, most probably attributable to vismodegib, or patient withdrawal of consent.
  Interventions: Drug: Vismodegib; Drug: Rosiglitazone
- Vismodegib + oral contraceptive (Experimental): Participants received the oral contraceptive norethindrone 1 mg/ethinyl estradiol 35 µg (Ortho-Novum 1/35®) orally on Days 1 and 8 of the study. Participants also received vismodegib 150 mg orally once a day beginning on Day 2 until one of the following occurred; disease progression, intolerable toxicity, most probably attributable to vismodegib, or patient withdrawal of consent.
  Interventions: Drug: Vismodegib; Drug: Norethindrone/ethinyl estradiol

INTERVENTIONS:
Drug: Vismodegib — Vismodegib was supplied in hard gelatin capsules.
  Other Names: GDC-0449
Drug: Rosiglitazone — Rosiglitazone was supplied in tablets.
  Arms: Vismodegib + rosiglitazone
Drug: Norethindrone/ethinyl estradiol — Norethindrone/ethinyl estradiol was supplied in tablets.
  Arms: Vismodegib + oral contraceptive

SUMMARY:
This is a single-arm, multicenter, Phase Ib study designed to describe the effect of GDC-0449 on the pharmacokinetics of rosiglitazone and oral contraceptives in patients with advanced solid tumors who are refractory to treatment or for whom no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of incurable, locally advanced, or metastatic solid malignancy that has failed to respond to at least one prior regimen or for which there is no standard therapy
* Documented negative serum pregnancy test for women of childbearing potential and use of two forms of contraception. Contraception must be used while the patient is enrolled in the study and for 12 months after the patient discontinues from the study.
* For men with female partners of childbearing potential, agreement to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 3 months after their last dose of GDC-0449.
* Agreement not to donate blood or blood products during the study and for at least 12 months after their last dose of GDC-0449
* For male patients, agreement not to donate sperm during the study and for at least 3 months after their last dose of GDC-0449
* Adequate hematopoietic capacity
* Adequate renal function
* Adequate hepatic function
* At least 3 weeks since the patient's last chemotherapy, investigational agent, radiation therapy, or major surgical procedure and recovery to pre-treatment baseline or stabilization of all treatment-related toxicities

Exclusion Criteria:

* Active infection requiring intravenous (IV) antibiotics
* Clinically important history of liver disease significantly impairing hepatic function, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Any medical condition or diagnosis that would likely impair absorption of an orally administered drug
* Pregnant or lactating
* Treatment with excluded medications, including strong CYP450 inhibitors and inducers, within 2 weeks of study entry
* Male patients already receiving rosiglitazone
* Male patients with a known contraindication to rosiglitazone
* Female patients already receiving oral contraception < 14 days prior to Day 1
* Female patients with known contraindication to oral contraceptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Colburn, Pharm.D., Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Stanford, California
  - Detroit, Michigan
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vismodegib + Rosiglitazone | Vismodegib + Oral Contraceptive
Started | 24 | 28
Completed | 5 | 8
Not Completed | 19 | 20
Not completed — Adverse Event | 2 | 1
Not completed — Death | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Disease progression | 11 | 16

BASELINE CHARACTERISTICS:
Population: Safety-evaluable population: All participants who received any amount of study drug (vismodegib or rosiglitazone or norethindrone/ethinyl estradiol).
Groups:
- Total: Total of all reporting groups
Arm/Group | Vismodegib + Rosiglitazone | Vismodegib + Oral Contraceptive | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (14.4) | 59.2 (14.6) | 60.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 27 | 27
  Male | 24 | 1 | 25

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio of the Area Under the Plasma Concentration-time Curve From 0 to Infinity (AUC[0-inf]) of Rosiglitazone
Description: On Days 1 and 8, blood samples were taken prior to the administration of rosiglitazone and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose. Plasma concentrations of rosiglitazone were determined using a validated liquid chromatography mass spectrometry/mass spectrometry (LC MS/MS) assay. Individual and mean plasma rosiglitazone concentration versus time data were tabulated and plotted by analyte. The pharmacokinetic parameters of each analyte were calculated using standard non-compartmental methods (WinNonlin version 5.2.1, Pharsight Corp., Mountain View, CA). The geometric mean ratio of AUC(0-inf) of rosiglitazone was defined as the AUC(0-inf) of rosiglitazone on Day 8/AUC(0-inf) of rosiglitazone on Day 1.
Time Frame: Pre-dose and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose
Population: Pharmacokinetic population: All participants with pharmacokinetic data on Day 1 and Day 8.
Measure: Number (90% Confidence Interval); unit: ng/mL*hr
Arm/Group | Vismodegib + Rosiglitazone
Number analyzed (Participants) | 24
ng/mL*hr | 92.0 [87.4 to 96.8]

2. Primary Outcome: Geometric Mean Ratio of the Maximum Plasma Concentration (Cmax) of Rosiglitazone
Description: On Days 1 and 8, blood samples were taken prior to the administration of rosiglitazone and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose. Plasma concentrations of rosiglitazone were determined using a validated liquid chromatography mass spectrometry/mass spectrometry (LC MS/MS) assay. Individual and mean plasma rosiglitazone concentration versus time data were tabulated and plotted by analyte. The pharmacokinetic parameters of each analyte were calculated using standard non-compartmental methods (WinNonlin version 5.2.1, Pharsight Corp., Mountain View, CA). The geometric mean ratio of Cmax of rosiglitazone was defined as the Cmax of rosiglitazone on Day 8/ Cmax of rosiglitazone on Day 1.
Time Frame: Pre-dose and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose
Population: Pharmacokinetic population: All participants with pharmacokinetic data on Day 1 and Day 8.
Measure: Number (90% Confidence Interval); unit: ng/mL
Arm/Group | Vismodegib + Rosiglitazone
Number analyzed (Participants) | 24
ng/mL | 93.1 [85.0 to 102]

3. Primary Outcome: Geometric Mean Ratio of the Area Under the Plasma Concentration-time Curve From 0 to Infinity (AUC[0-inf]) of Ethinyl Estradiol and Norethindrone
Description: On Days 1 and 8, blood samples were taken prior to the administration of the contraceptive norethindrone 1 mg/ethinyl estradiol 35 µg (Ortho-Novum 1/35®) and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose. Plasma concentrations of ethinyl estradiol and norethindrone were determined using a validated liquid chromatography mass spectrometry/mass spectrometry (LC MS/MS) assay. Individual and mean plasma ethinyl estradiol and norethindrone concentration versus time data were tabulated and plotted by analyte. The pharmacokinetic parameters of each analyte were calculated using standard non-compartmental methods (WinNonlin version 5.2.1, Pharsight Corp., Mountain View, CA). The geometric mean ratios of AUC(0-inf) of ethinyl estradiol and norethindrone were defined as the ratios of AUC(0-inf) of ethinyl estradiol and norethindrone on Day 8 divided by AUC(0-inf) of ethinyl estradiol and norethindrone on Day 1, respectively.
Time Frame: Pre-dose and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose
Population: Pharmacokinetic population: All participants with pharmacokinetic data on Day 1 and Day 8.
Measure: Number (90% Confidence Interval); unit: ng/mL*hr
Arm/Group | Vismodegib + Oral Contraceptive
Number analyzed (Participants) | 27
ng/mL*hr
  Ethinyl estradiol | 99.6 [92.9 to 107]
  Norethindrone | 123 [115 to 131]

4. Primary Outcome: Geometric Mean Ratio of the Maximum Plasma Concentration (Cmax) of Ethinyl Estradiol and Norethindrone
Description: On Days 1 and 8, blood samples were taken prior to the administration of the contraceptive norethindrone 1 mg/ethinyl estradiol 35 µg (Ortho-Novum 1/35®) and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose. Plasma concentrations of ethinyl estradiol and norethindrone were determined using a validated liquid chromatography mass spectrometry/mass spectrometry (LC MS/MS) assay. Individual and mean plasma ethinyl estradiol and norethindrone concentration versus time data were tabulated and plotted by analyte. The pharmacokinetic parameters of each analyte were calculated using standard non-compartmental methods (WinNonlin version 5.2.1, Pharsight Corp., Mountain View, CA). The geometric mean ratios of Cmax of ethinyl estradiol and norethindrone were defined as the ratios of Cmax of ethinyl estradiol and norethindrone on Day 8 divided by Cmax of ethinyl estradiol and norethindrone on Day 1, respectively.
Time Frame: Pre-dose and 30 minutes, and 1, 2, 3, 4, and 6 hours, between 8 and 12 hours, and 24 hours post-dose
Population: Pharmacokinetic population: All participants with pharmacokinetic data on Day 1 and Day 8.
Measure: Number (90% Confidence Interval); unit: ng/mL
Arm/Group | Vismodegib + Oral Contraceptive
Number analyzed (Participants) | 27
ng/mL
  Ethinyl estradiol | 105 [94.4 to 116]
  Norethindrone | 112 [101 to 124]

ADVERSE EVENTS:
Description: Safety-evaluable population: All participants who received any amount of study drug (vismodegib or rosiglitazone or norethindrone/ethinyl estradiol).
Arm/Group | Vismodegib + Rosiglitazone | Vismodegib + Oral Contraceptive
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 22/24 | 20/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib + Rosiglitazone (N=24) | Vismodegib + Oral Contraceptive (N=28)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 4 | 8
Vomiting (Gastrointestinal disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 9 | 9
Headache (Nervous system disorders) | 3 | 1
Hypogeusia (Nervous system disorders) | 2 | 0
Fatigue (General disorders) | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Weight decreased (Investigations) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.